CLINICAL TRIAL: NCT03663452
Title: Targeted Strategies to Accelerate Evidence-Based Psychotherapy (EBP) Implementation in Military Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Palo Alto Veterans Institute for Research (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Carmen McLean, Co-Principal Investigator, Palo Alto Veterans Institute for Research
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: ROS0029
Record Dates: First submitted 2018-09-04; First posted 2018-09-10 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: This project will use a cluster-randomized stepped wedge design in eight MHS behavioral health outpatient clinics. All sites first receive PE training, and are randomly allocated to receive the TACTICS intervention either 5, 10, or 15 months later.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prolonged exposure training (Active Comparator)
  Interventions: Behavioral: Prolonged exposure training
- TACTICS (Experimental)
  Interventions: Behavioral: Targeted Assessment and Context-Tailored Implementation of Change Strategies (TACTICS)

INTERVENTIONS:
Behavioral: Targeted Assessment and Context-Tailored Implementation of Change Strategies (TACTICS) — TACTICS begins with a mixed methods assessment (using data from medical records, staff surveys, and staff interviews) to identify barriers and facilitators of PE use in each clinic. From a menu of implementation strategies that can be matched to local conditions, an implementation plan is developed in collaboration with clinic personnel and deployed to address specific barriers and leverage strengths at each clinic site over a 5-month period.
  Arms: TACTICS
Behavioral: Prolonged exposure training — Providers will receive a 2-day workshop training in the delivery of prolonged exposure, followed by weekly phone clinical consultation.
  Arms: Prolonged exposure training

SUMMARY:
This study will evaluate a program designed to increase military treatment facilities' use of Prolonged Exposure (PE), an evidence-based psychotherapy for PTSD. The results will determine whether this program increases PE use and improves patient outcomes compared to conventional provider training in PE, and feedback from clinic leaders and staff will be used to gauge program usability, identify successful components, and refine program for expansion.

DETAILED DESCRIPTION:
Background: Posttraumatic stress disorder (PTSD) is a significant problem in the military, impacting as many as 1 in 5 military personnel. Efforts to disseminate evidence-based treatments for PTSD such as Prolonged Exposure (PE) therapy throughout the Military Health System (MHS) have relied primarily on provider training. These have yielded mixed results, because they do not directly address barriers that may prevent providers from using a new treatment after they gave been trained in it. Barriers to using PE within the MHS are complex and exist at various levels of organization from the provider level to the "outer context" (i.e., higher headquarter policies, guidelines). In addition, barriers may vary considerably from one military treatment facility to another. Thus, implementation strategies to improve use of PE need to be tailored to conditions in each clinic site.

Objectives: The primary objective is to develop and implement a novel approach, Targeted Assessment and Context-Tailored Implementation of Change Strategies (TACTICS), to improve the implementation of PE and to test its impact on care over and above clinician training only. TACTICS provides a menu of implementation strategies that can be matched to local conditions. These strategies are informed by the implementation science literature and by prior experience working with military clinics, The TACTICS process begins with a mixed methods assessment (using data from medical records, staff surveys, and staff interviews) to identify barriers and facilitators of PE use in each clinic. Implementation strategies are then selected in collaboration with clinic personnel and deployed to address specific barriers and leverage strengths at each clinic site.

Specific Aims: 1) To examine the impact of a multi-modal, tailored approach (TACTICS) over and above conventional PE training on the proportion of PTSD patients who receive PE for PTSD, as measured by Natural Language Processing (NLP) of psychotherapy progress notes (primary measure) and clinician-selected psychotherapy modality (secondary measure). 2) To examine the impact of TACTICS over and above conventional PE training on mean improvement in Military Treatment Facility (MTF) clinic patients' scores on the PTSD Checklist (PCL) for DSM-5 (fifth edition of the Diagnostic and Statistical Manual of Mental Disorders, PCL-5). 3) To evaluate the usability of and overall satisfaction with TACTICS among senior leaders, clinic leaders, and providers, as assessed by qualitative data obtained from the post-TACTICS feedback interviews. The study will also aim to identify TACTICS components that a) were seen as most useful by participants and appear to contribute to implementation success; b) are potentially helpful but require modifications; and c) are potentially unnecessary and do not appear to contribute to implementation success. Exploratory aims include: A) To assess the impact of TACTICS (over and above PE training) on provider and clinic-level factors theorized to facilitate implementation in the Consolidated Framework for Implementation Research (CFIR). These proximal factors include changes in provider knowledge/beliefs about PE, provider self-efficacy, burnout, implementation climate, and leadership engagement, as assessed through online surveys. B) To explore whether changes in additional CFIR-theorized provider- and clinic-level factors (based on emergent themes in qualitative needs assessment interviews and exit interviews) are associated with greater improvements in reach (i.e., a greater number of patients receiving PE) and effectiveness (i.e., greater improvement in PTSD symptoms as measured by the PCL-5). C) To examine the TACTICS implementation strategies employed at each site in connection with increase in PE receipt, to determine whether any particular strategies had a positive or negative impact on PE receipt. D) To evaluate the impact of TACTICS over and above conventional PE training on self-reported levels of PE fidelity, as measured by NLP data of psychotherapy progress notes. E) To examine patient characteristics (e.g., depression, generalized anxiety, recent hospitalizations, other psychiatric diagnoses) that may be associated with PE receipt.

Study Design. This project will use a cluster-randomized stepped wedge design in eight MHS behavioral health outpatient clinics. Randomization will occur at the clinic level to account for the clustering of providers within clinics. All clinics receive the whole intervention package, but timing is randomly assigned. Participants will include the behavioral health providers and relevant clinic and hospital leadership. During a baseline phase, provider training in PE will be delivered. During the second phase, a clinic-based needs assessment will be conducted followed by the implement of TACTICS components. Selection of implementation strategies will be guided by the results of the needs assessments and well-established implementation science frameworks. Results of the second phase will determine the impact of TACTICS over and above clinician training.

Significance. Accelerating the use of PE for PTSD within the MHS will increase the number of service members in need who can access, and hopefully benefit, from an effective PTSD treatment. In turn, as more patients recover successfully, behavioral health clinic capacity will increase and more service members will receive care. The project will identify solutions for the unique challenges to implementation of PE in the MHS, and, if effective, TACTICS may represent a scalable approach to accelerating the use of other behavioral health best practices in military settings

ELIGIBILITY:
Inclusion Criteria:

* Provides behavioral health care to PTSD patients

Exclusion Criteria:

* Plans to relocate within next 5 months

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
PE use | Baseline to 20 months
  The proportion of PTSD patients who receive PE, as measured by coded electronic medical record data

SECONDARY OUTCOMES:
Change in patients' PTSD severity | Baseline to 20 months
  Patients' PTSD symptoms, as measured by change on a PTSD symptom measure routinely collected at behavioral health appointments.

OTHER OUTCOMES:
TACTICS usability and satisfaction | Immediately after the 5-month TACTICS intervention
  Usability of and overall satisfaction with TACTICS among senior leaders, clinic leaders, and providers, as assessed through post-TACTICS qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen McLean, PhD, Principal Investigator — carmen.mclean4@va.gov
Locations (8):
- United States (8):
  - Bassett Army Community Hospital / Ft. Wainwright, Fairbanks, Alaska
  - Mental Health Clinic / Travis Air Force Base, Fairfield, California
  - Naval Hospital Jacksonville / Naval Air Station Jacksonville, Jacksonville, Florida
  - Blanchfield Army Community Hospital (BACH) / Fort Campbell, Fort Campbell North, Kentucky
  - 81st Medical Group / Keesler Air Force Base, Biloxi, Mississippi
  - 49th Medical Group / Holloman Air Force Base, Alamogordo, New Mexico
  - William Beaumont Army Medical Center (WBAMC) / Fort Bliss, El Paso, Texas
  - Brooke Army Medical Center (BAMC) / Fort Sam Houston, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rosen CS, Davis CA, Riggs D, Cook J, Peterson AL, Young-McCaughan S, Comtois KA, Haddock CK, Borah EV, Dondanville KA, Finley EP, Jahnke SA, Poston WSC, Wiltsey-Stirman S, Neitzer A, Broussard CR, Brzuchalski MA, Clayton MSP, Conforte LAM, Flores A, Hein J, Keith CF, Jinkerson CJ, Letendre M, Nofziger D, Pollick K, Santiago CK, Waggoner LCJ, Woodworth C, McLean CP; TACTICS Research Group. Targeted Assessment and Context-Tailored Implementation of Change Strategies (TACTICS) to increase evidence based psychotherapy in military behavioral health clinics: Design of a cluster-randomized stepped-wedge implementation study. Contemp Clin Trials. 2020 Jun;93:106008. doi: 10.1016/j.cct.2020.106008. Epub 2020 Apr 21. PMID 32330670